CLINICAL TRIAL: NCT07070141
Title: Bruxism and Temporomandibular Joint Vibrational Patterns: Insights From Joint Vibration Analysis
Brief Title: Bruxism and Temporomandibular Joint Vibrational Analysis Study
Acronym: BRUX-TMJ
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Serdar Gozler, ass. prof, Atlas University
Other Study IDs: 2024-ATLAS-MSEHF-002
Record Dates: First submitted 2025-06-25; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Bruxism; Temporomandibular Disorder (TMD)
Keywords: Bruxism; Joint Vibration analysis; Sound frequencies; Temporomandibular,; Temporomandibular joint
MeSH Terms: conditions — Bruxism; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy
  Interventions: Diagnostic Test: Diagnostic work up
- bruxism: self-reported bruxism
  Interventions: Diagnostic Test: Diagnostic work up

INTERVENTIONS:
Diagnostic Test: Diagnostic work up — None intervention

SUMMARY:
Background and Rationale

Bruxism is a repetitive jaw-muscle activity involving clenching or grinding of the teeth. Although its pathophysiology remains unclear, it is hypothesized that bruxism may contribute to biomechanical alterations in the temporomandibular joint (TMJ). Joint Vibration Analysis (JVA) is a non-invasive method capable of detecting vibrational patterns associated with TMJ function. This study protocol aims to assess the potential association between bruxism and TMJ vibrational characteristics in adults.

Objectives

The primary objective is to determine whether there is a difference in TMJ vibrational parameters between individuals with clinically diagnosed bruxism and individuals without signs or symptoms of bruxism. The secondary objective is to explore the relationship between bruxism severity and specific vibrational parameters measured by JVA.

Study Design

This is a retrospective observational study of patient records collected between January 2020 and May 2025 at the Istanbul Atlas University TMD Clinic.

Study Population

* Inclusion Criteria:
* Adults aged 18-45 years
* Documented bruxism evaluation
* Complete Joint Vibration Analysis (JVA) recordings
* Exclusion Criteria:
* History of orthodontic treatment within the past year
* TMJ surgery or major facial trauma
* Neurological or systemic inflammatory conditions
* Pregnancy at time of evaluation
* Use of medications affecting neuromuscular activity

Sample Size

Approximately 195 patient records meeting eligibility criteria will be analyzed. The bruxism group is expected to include ~175 participants, and the control group ~20 participants.

Methodology

Clinical data include patient-reported bruxism history, maximum mouth opening measurements, and TMJ clinical assessments. JVA recordings will be used to obtain vibrational parameters such as peak frequency, median frequency, amplitude, and total vibrational energy. Standardized protocols for JVA will be applied to all included patients.

Statistical Analysis

Data normality will be assessed. For normally distributed variables, independent t-tests will be used to compare groups; for non-normally distributed variables, Mann-Whitney U tests will be applied. Correlation between bruxism severity and vibrational parameters will be evaluated using Spearman's rank correlation. Multiple linear regression may be used to analyze the predictive value of bruxism indicators.

Ethics

The study protocol has been approved by the Istanbul Atlas University Clinical Research Ethics Committee (Approval No: E-22686390-050.99-66516). Informed consent for use of anonymized data was obtained at the time of clinical examination.

DETAILED DESCRIPTION:
Bruxism involves repetitive jaw-muscle activity, including clenching and grinding, which may generate excessive and chronic mechanical loading on the temporomandibular joint (TMJ). Although its causal link to TMJ disorders is still debated, it is hypothesized that bruxism-induced stress may lead to internal joint changes, detectable as vibrational anomalies.

Joint Vibration Analysis (JVA) is a non-invasive, real-time diagnostic modality that records vibrational events within the TMJ during mandibular movements. By analyzing parameters such as peak frequency (Hz), median frequency (Hz), amplitude (µV), and total energy (Pa·s), JVA enables objective assessment of intra-articular mechanical behavior. These metrics help differentiate between normal joint function and pathological conditions such as disc displacement or degenerative changes.

This retrospective observational study will assess whether individuals with clinically identified bruxism exhibit distinct vibrational profiles compared to asymptomatic controls. Patient records collected at the Istanbul Atlas University TMD Clinic between January 2020 and May 2025 will be included. Bruxism classification will be based on a standardized clinical scale, incorporating both self-reported symptoms (e.g., morning jaw fatigue, tooth wear, headache) and clinical signs (e.g., hypertrophic masseter muscles, linea alba, occlusal facets).

JVA recordings will be obtained using the BioJVA™ system (BioResearch Associates, Inc.), following a uniform protocol: bilateral sensor placement over the TMJs, seated posture with back support, and execution of five maximal open-close mandibular cycles. Calibration procedures will ensure data consistency across sessions. Demographic data (age, gender), maximum mouth opening (MMO), presence of joint sounds (clicks, crepitus), and JVA output parameters will be recorded.

Statistical analysis will include comparative tests (e.g., t-test, Mann-Whitney U) between bruxism and control groups, and correlation analyses (e.g., Pearson or Spearman coefficients) between vibrational variables and bruxism severity scores. Multivariate models may be used to control for age and gender effects.

This study protocol is ethically approved by the Istanbul Atlas University Clinical Research Ethics Committee. Anonymized data from consenting patients will be used in compliance with institutional and international research standards.

Findings from this research are expected to clarify the biomechanical effects of bruxism on TMJ structures and support the utility of JVA as an objective adjunct tool in the functional evaluation of temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 45 years
* Patients treated at the specialized TMD Clinic of Istanbul Atlas University
* Presence of at least one diagnostic criterion (e.g., orofacial pain, joint clicking, limited mandibular movement)

Exclusion Criteria:

* Patients with incomplete clinical documentation
* Individuals with systemic diseases affecting joint or muscle function
* Patients with a history of maxillofacial trauma or surgery
* Patients outside the specified age range

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bruxism
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Peak frequency of TMJ sounds | Baseline (single assessment at initial visit)
  Peak frequency refers to the dominant frequency component in the TMJ sound spectrum, measured during jaw opening. Unit of Measure: Hz

SECONDARY OUTCOMES:
Presence and severity of bruxism symptoms based on clinical assessment | Baseline
  Bruxism symptoms (such as tooth wear, muscle pain, or jaw fatigue) are assessed during clinical examination and rated using a standard severity scale. Unit of Measure: Binary (Yes/No) and clinical scale (e.g., 0-3 severity index)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Kâğıthane, Istanbul, Turkey (Türkiye)